CLINICAL TRIAL: NCT06490172
Title: The Effects of Extracorporeal Shock Wave Therapy as a Treatment Intervention for Chronic Adhesive Capsulitis: a Mixed Methods Pilot Study
Brief Title: Shock Wave Therapy as a Treatment Intervention for Frozen Shoulder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Stirling (Other)
Responsible Party: Principal Investigator, Crystal Reno, Professional Clinical Doctorate Student, University of Stirling
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 18192
Record Dates: First submitted 2024-03-11; First posted 2024-07-08 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Shoulder Pain; Adhesive Capsulitis of Shoulder
Keywords: shock wave therapy; frozen shoulder; adhesive capsulitis; shoulder pain; physiotherapy; lithotripsy
MeSH Terms: conditions — Shoulder Pain; Bursitis | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Intervention Model Description: Mixed Methods Explanatory Sequential Design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Delphi Study (No Intervention): The survey will be re-circulated a minimum of three, and maximum of four rounds, with an aim for a minimum of 20 participants and response rate of greater than 70 percent per round. The results will be collected and collated at each round to determine a consensus amongst shoulder specialists for further review. This information will be used to guide the treatment protocol in phase two.
- Shock wave therapy quantitative data collection and analysis (Experimental): This phase will involve the piloting of the shock wave therapy protocol determined by the results collected in phase one Delphi study
  Following participant consent, the research healthcare practitioner will provide patient reported outcome measure questionnaires for the participant to complete independently to measure baseline data. This will occur at baseline, 6 and 12 weeks following shock wave therapy treatment.
  Interventions: Device: Shock wave therapy
- Qualitative semi-structured interviews (No Intervention): All participants in phase 2 and those who declined participation in the quantitative study at the recruitment stage will be invited to take part in semi-structured qualitative interviews of a duration of 30 - 45 minutes. The interview protocol and questions will be developed based on the findings of the quantitative data analysis. Interviews will take place approximately 12 weeks from last ESWT treatment.

INTERVENTIONS:
Device: Shock wave therapy — Radial Extracorporeal Shock Wave Therapy and feasibility as treatment for adhesive capsulitis
  Arms: Shock wave therapy quantitative data collection and analysis

SUMMARY:
Adhesive capsulitis (AC) is a debilitating condition that causes global restriction and pain at the glenohumeral joint. Physiotherapy treatment is often first line treatment management. Patients with failed conservative management are commonly referred to a specialist consultant for further treatment. Over the last 20 years, extracorporeal shock wave therapy (ESWT) has gained popularity as a treatment for various orthopaedic presentations, including chronic soft tissue conditions, being non-invasive, resulting in good outcomes with minimal side effects. There is a lack of evidence on the clinical effectiveness of ESWT for chronic AC following failed conservative treatments, with the available literature reporting positive outcomes, however, with heterogeneity in treatment protocols. This proposed study aims to explore the feasibility of a full trial of ESWT as a treatment for AC using a standardised treatment protocol, and clinical effects on outcomes of pain, function and shoulder joint range of movement in persons with chronic adhesive capsulitis.

A Delphi study will first explore expert opinion for the optimum treatment protocol of ESWT as a treatment for chronic AC, followed by a mixed methods explanatory sequential study that includes a pilot trial with nested qualitative interviews. The Shoulder Pain and Disability Index, numerical pain rating scale, EuroQol-5D, and digital goniometer will be used to measure self-reported pain and function, pain, health-related quality of life, and shoulder joint range of movement, respectively. Quantitative data will be analysed by descriptive statistics. Qualitative data will be collected through semi-structured interviews. Interview data will be analysed using Braun and Clarke's inductive thematic analysis approach. The study will be conducted in an out-patient clinical setting in a community health hub facility, with patients recruited from an NHS Orthopaedics waitlist. Data collection is planned over a nine month period. This study is not affiliated with funding streams.

DETAILED DESCRIPTION:
Shoulder AC, commonly known as frozen shoulder, is a self-limiting condition that affects three to five percent of the population and up to 20 to 30 percent in persons with diabetes mellitus. Its aetiology is still being understood with evidence supporting a chronic state of low-grade inflammation and elevation of pro-inflammatory lipoproteins resulting in fibrotic changes in the glenohumeral capsule. This results in pain, reduced shoulder range of movement (ROM) and functional disability that can spontaneously resolve between one to three years, with 40 percent reporting persistent symptoms at long-term follow up (mean follow up time 4.4 years, range 2 - 20 years). AC can occur spontaneously, as a primary insidious onset, or secondary, following a post-traumatic event such as shoulder surgery or rotator cuff injury. Treatment for AC commonly consists of conservative management interventions including pharmacotherapy, physiotherapy, and corticosteroid injection, with referral to secondary care if symptoms persist for interventions such as manipulation under anaesthesia and arthroscopic capsular release.

The treatment interventions or surgical procedures for AC may not always be effective or suitable for all patients due to conditions that may increase risk of complications such as respiratory conditions, allergies, previous surgery complications, co-morbidities (e.g., liver, cardiovascular and kidney disease), and patient choice. Untreated conditions and long-wait times can lead to chronicity further impacting an individual's health and increasing costs to the National Health Service (NHS). Musculoskeletal (MSK) conditions are estimated to cost to the British government an estimated £7 billion per year, accounting for one third of the NHS budget. In a United Kingdom (UK) health survey evaluating the prevalence of chronic pain (duration of pain 12 weeks or more), labelled MSK conditions as a long-lasting illness, accounting for 81 percent of participants, and of this, 24 percent involving the shoulder. Chronic MSK pain has also been linked to 17.5 percent of work absences, anxiety, depression, and health inequalities.

Over the last 20 years, EWST, has gained popularity as a treatment modality for orthopaedics conditions such as chronic tendinopathies. EWST can be generated as focused high- energy (>0.60 millijoules (mj)/mm2) shock waves or emitted as radial low (<0.08 mJ/mm2) to medium-energy (<0.28 mJ/mm2) shock waves. ESWT stimulates soft tissue healing via a biological response of mechanotransduction through neovascularisation, reduction of tendon matrix inflammatory markers such as metalloproteinases and interleukins, assists with the migration and differentiation of mesenchymal stem cells, and enhances the natural healing microenvironment. To date, therapeutic EWST has been shown to be clinically effective to treat bone non-unions, chronic soft tissue disorders such as tendinopathies and recalcitrant MSK conditions commonly involving the supraspinatus muscle tendon, patellar tendon, Achilles tendon and plantar fascia, and has become a favourable alternative treatment for individuals who have exhausted conventional conservative interventions.

A review of the literature exploring the use of ESWT as a treatment for chronic AC found seven randomised control trials (RCT) reporting significant improvements in function, pain and shoulder ROM in groups that received ESWT. The literature found improvements in all outcomes within 12 weeks when compared to a control group.

Although the literature demonstrates positive outcomes, due to the small number of studies, small sample sizes, and heterogeneity of treatment protocols, there is insufficient evidence for it to be a recommended treatment for AC by national health guidelines (e.g., National Institute for Health and Care Excellence). Further research is therefore required to determine the acceptability and viability of this intervention in the UK healthcare framework, with potential to conduct a full-scale RCT.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged 18 years and older.
2. Diagnosis of primary or secondary shoulder AC of a greater than three-month duration.
3. Diagnosis of AC by an orthopaedic consultant or upper limb Advanced Practice Physiotherapist.
4. Participants can attend an outpatient rural physiotherapy department to receive shockwave therapy intervention.
5. They understand English.

Exclusion Criteria:

1. Participants who have bilateral shoulder pain, capsular tightness, calcific rotator cuff tendinitis, rotator cuff tear (atraumatic or traumatic), previous surgery on the affected shoulder, shoulder fracture, dislocation or subluxation, glenohumeral or acromioclavicular arthritis, malignancy, inflammatory disorders, neuromuscular disorders, presence of severe osteoporosis, pulmonary diseases, implanted pacemaker and pregnancy.
2. They have conditions related to ESWT contraindications (e.g., pregnancy, pacemaker, metal work or joint replacement near the treatment site, blood clotting disorder, use of anti-coagulants, less than six weeks of receiving a steroid injection over treatment site, malignancy, local infection or open wounds, skeletal growth places, under 18 years old).
3. Symptom duration less than 12 weeks.
4. Absent or altered skin sensation.
5. They are unable to give full informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Recruitment and rejection rate | 18 months
  Estimate the proportion of patients screened who meet the eligibility criteria. This will be analysed with descriptive statistics using IBM SPSS Statistical Software. This will be displayed as a numerical value with standard deviation
Retention rate | 18 month
  Adherence and compliance to intervention and home exercise programme, follow-up and drops out. This will be analysed with descriptive statistics using IBM SPSS Statistical Software. This will be displayed as a numerical value with standard deviation

SECONDARY OUTCOMES:
The Shoulder Pain and Disability Index | 0, 6, and 12 weeks.
  Self-reported pain and function in shoulder conditions. 13 item questionnaire that assesses two domains, pain and disability, that best represents their shoulder symptoms over a week. The scale is scored from a zero, 'no pain / no difficulty,' to 10, 'worst pain imaginable / so difficult requires help', with higher scores indicating increase impairment or disability, and can be used to monitor change over time. A difference of eight points is the minimal detectable change for clinical significance.
Numerical Pain Rating Scale | 0, 6, and 12 weeks.
  One-dimensional tool used to measure pain both at rest and during movement. It is a 11-point scale for self-reported pain, zero meaning 'no pain' to 10 'extreme pain / worse pain possible,' at the time the questionnaire is administered and has been found to be more versatile being delivered in both verbal and written formats. Minimal clinical difference of change sore for general conditions is 3.0cm, and rotator cuff pain is 1.4cm on scale.
EuroQoL-5D-5L | 0, 6, and 12 weeks.
  Questionnaire measuring health-related quality of life. It measures five dimensions of health, mobility, self-care, usual activities, pain and discomfort, and anxiety and depression, on a five-level scale. A score of one across all five categories represents the best possible health, whereas a score of five across all five categories represents the worst health status. The EQ-5D-5L also includes a perceived health status demonstrated as a visual analogue scale with grade ranging from zero, the worst possible health status, to 100, the best possible health status.
Digital Goniometry | 0, 6, and 12 weeks.
  A digital goniometer or smart phone application digital inclinometer will be used to measure shoulder joint passive ROM.

CONTACTS AND LOCATIONS:
Overall Officials: Crystal Reno, Principal Investigator — University of Stirling

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zreik NH, Malik RA, Charalambous CP. Adhesive capsulitis of the shoulder and diabetes: a meta-analysis of prevalence. Muscles Ligaments Tendons J. 2016 May 19;6(1):26-34. doi: 10.11138/mltj/2016.6.1.026. eCollection 2016 Jan-Mar. PMID 27331029
- [Background] Le HV, Lee SJ, Nazarian A, Rodriguez EK. Adhesive capsulitis of the shoulder: review of pathophysiology and current clinical treatments. Shoulder Elbow. 2017 Apr;9(2):75-84. doi: 10.1177/1758573216676786. Epub 2016 Nov 7. PMID 28405218
- [Background] Kraal T, Lubbers J, van den Bekerom MPJ, Alessie J, van Kooyk Y, Eygendaal D, Koorevaar RCT. The puzzling pathophysiology of frozen shoulders - a scoping review. J Exp Orthop. 2020 Nov 18;7(1):91. doi: 10.1186/s40634-020-00307-w. PMID 33205235
- [Background] Hand C, Clipsham K, Rees JL, Carr AJ. Long-term outcome of frozen shoulder. J Shoulder Elbow Surg. 2008 Mar-Apr;17(2):231-6. doi: 10.1016/j.jse.2007.05.009. Epub 2007 Nov 12. PMID 17993282
- [Background] NICE (2017) Scenario: frozen shoulder. Available: https://cks.nice.org.uk/topics/shoulder-pain/management/frozen-shoulder/ [Accessed: 04 November 2022].
- [Background] Dennis, L., Brealey, S., Rangan, A., Rookmoneea, M. and Watson, J. (2010) Managing idiopathic frozen shoulder: a survey of health professionals' current practice and research priorities. Shoulder and Elbow, 2 (4), pp. 294-300.
- [Background] Smith G, D'Cruz JR, Rondeau B, Goldman J. General Anesthesia for Surgeons. 2023 Aug 5. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK493199/ PMID 29630251
- [Background] Wang CJ. Extracorporeal shockwave therapy in musculoskeletal disorders. J Orthop Surg Res. 2012 Mar 20;7:11. doi: 10.1186/1749-799X-7-11. PMID 22433113
- [Background] Taylor J, Dunkerley S, Silver D, Redfern A, Talbot N, Sharpe I, Guyver P. Extracorporeal shockwave therapy (ESWT) for refractory Achilles tendinopathy: A prospective audit with 2-year follow up. Foot (Edinb). 2016 Mar;26:23-9. doi: 10.1016/j.foot.2015.08.007. Epub 2015 Aug 31. PMID 26802946
- [Background] Lohrer H, Nauck T, Dorn-Lange NV, Scholl J, Vester JC. Comparison of radial versus focused extracorporeal shock waves in plantar fasciitis using functional measures. Foot Ankle Int. 2010 Jan;31(1):1-9. doi: 10.3113/FAI.2010.0001. PMID 20067715
- [Background] Waugh CM, Morrissey D, Jones E, Riley GP, Langberg H, Screen HR. In vivo biological response to extracorporeal shockwave therapy in human tendinopathy. Eur Cell Mater. 2015 May 15;29:268-80; discussion 280. doi: 10.22203/ecm.v029a20. PMID 25978115
- [Background] Chen CY, Hu CC, Weng PW, Huang YM, Chiang CJ, Chen CH, Tsuang YH, Yang RS, Sun JS, Cheng CK. Extracorporeal shockwave therapy improves short-term functional outcomes of shoulder adhesive capsulitis. J Shoulder Elbow Surg. 2014 Dec;23(12):1843-1851. doi: 10.1016/j.jse.2014.08.010. PMID 25441567
- [Background] El Naggar TEDM, Maaty AIE, Mohamed AE. Effectiveness of radial extracorporeal shock-wave therapy versus ultrasound-guided low-dose intra-articular steroid injection in improving shoulder pain, function, and range of motion in diabetic patients with shoulder adhesive capsulitis. J Shoulder Elbow Surg. 2020 Jul;29(7):1300-1309. doi: 10.1016/j.jse.2020.03.005. PMID 32553435
- [Background] Hameedi, I.A., Shadmehr, A., Malmir, K., Fereydounnia, S. and Shiravi, Z. (2022) Comparison of application of the radial vs. focused probes of extracorporeal shockwave therapy on pain, range of motion and function in patients with adhesive capsulitis. NeuroQuantology, 20 (6), pp. 2726.
- [Background] Hussein, A.Z. and Donatelli, R.A. (2016) The efficacy of radial extracorporeal shockwave therapy in shoulder adhesive capsulitis: a prospective, randomised, double-blind, placebo-controlled, clinical study. European Journal of Physiotherapy, 18 (1), pp. 63-76.
- [Background] Lee S, Lee S, Jeong M, Oh H, Lee K. The effects of extracorporeal shock wave therapy on pain and range of motion in patients with adhesive capsulitis. J Phys Ther Sci. 2017 Nov;29(11):1907-1909. doi: 10.1589/jpts.29.1907. Epub 2017 Nov 24. PMID 29200621
- [Background] Saldiran TC, Yazgan P, Akgol AC, Mutluay FK. Radial shock-wave therapy for frozen shoulder patients with type 2 diabetes mellitus: a pilot trial comparing two different energy levels. Eur J Phys Rehabil Med. 2022 Jun;58(3):412-422. doi: 10.23736/S1973-9087.22.07087-3. Epub 2022 Feb 22. PMID 35191654
- [Background] Vahdatpour B, Taheri P, Zade AZ, Moradian S. Efficacy of extracorporeal shockwave therapy in frozen shoulder. Int J Prev Med. 2014 Jul;5(7):875-81. PMID 25104999
- [Background] Eubank BH, Mohtadi NG, Lafave MR, Wiley JP, Bois AJ, Boorman RS, Sheps DM. Using the modified Delphi method to establish clinical consensus for the diagnosis and treatment of patients with rotator cuff pathology. BMC Med Res Methodol. 2016 May 20;16:56. doi: 10.1186/s12874-016-0165-8. PMID 27206853
- [Background] Eldridge SM, Chan CL, Campbell MJ, Bond CM, Hopewell S, Thabane L, Lancaster GA; PAFS consensus group. CONSORT 2010 statement: extension to randomised pilot and feasibility trials. BMJ. 2016 Oct 24;355:i5239. doi: 10.1136/bmj.i5239. PMID 27777223
- [Background] Lewis M, Bromley K, Sutton CJ, McCray G, Myers HL, Lancaster GA. Determining sample size for progression criteria for pragmatic pilot RCTs: the hypothesis test strikes back! Pilot Feasibility Stud. 2021 Feb 3;7(1):40. doi: 10.1186/s40814-021-00770-x. PMID 33536076
- [Background] Julious, S.A. (2005) Sample size of 12 per group rule of thumb for a pilot study. Pharmaceutical Statistics, 4 (4), pp. 287-291.
- [Background] Creswell, J. and Plano Clark, V. (2011) Designing and conducting mixed methods research. 2nd ed. Thousand Oaks, California: Sage Publications. Available: https://www.vlebooks.com/vleweb/product/openreader?id=none&isbn=9781412993654&uid=none
- [Background] Creswell, J. (2014) Research design. 4th ed. Thousand Oaks, California: SAGE Publications.
- [Background] EMS - Dolorclast (2021) Guided dolarclast therapy. Available: https://www.ems-dolorclast.com/sites/default/files/2021-11/FA-720_EN_Rev_B_GDT%20Sales%20Aid_Ed_07-2021_Light%20%281%29.pdf [Accessed: 09 February 2024].
- [Background] PHE (2019) Musculoskeletal health: a 5 year strategic framework for prevention across the lifecourse. London: Public Health England (PHE). Available: https://assets.publishing.service.gov.uk/government/uploads/system/uploads/attachment_data/file/810348/Musculoskeletal_Health_5_year_strategy.pdf [Accessed: 15 December 2022].
- [Background] PHE (2017) Chronic pain in adults 2017: health survey for england. Available: https://assets.publishing.service.gov.uk/government/uploads/system/uploads/attachment_data/file/940858/Chronic_Pain_Report.pdf [Accessed: 04 November 2022].
- [Background] OHID (2022) Musculoskeletal health: applying All Our Health. Available: https://www.gov.uk/government/publications/musculoskeletal-health-applying-all-our-health/musculoskeletal-health-applying-all-our-health#fn:1 [Accessed: 08 November 2022].
- [Background] Versus Arthritis (2021) The state of musculoskeletal health 2021: arthritis and other musculoskeletal conditions in numbers. Available: https://www.versusarthritis.org/media/24653/state-of-msk-health2-2021.pdf [Accessed: 15 November 2022].